CLINICAL TRIAL: NCT00661128
Title: Evaluating the Genetic Factors That May Lead to Sudden Cardiac Arrest (The GenSCA Study)
Brief Title: Genomics of Sudden Cardiac Arrest
Acronym: GenSCA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); King County Emergency Medical Services (Unknown); University of California, San Francisco (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Nona Sotoodehnia, Associate Professor of Medicine, Medicine/Cardiology, University of Washington
Other Study IDs: 35496; 1R01HL088456 (NIH)
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Death, Sudden, Cardiac
Keywords: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — De-identified white blood cells, red blood cells, plasma, and DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: European American people who have experienced SCA.
- 2: European American people who have not experienced SCA.
- 3: African American people who have experienced SCA.
- 4: African American people who have not experienced SCA.

SUMMARY:
Sudden cardiac arrest (SCA) is a sudden, unexpected loss of heart function. It is a leading cause of death, and more than 400,000 people in the United States die each year as a result of SCA. This study will analyze genetic samples of people who have experienced SCA and people who have not experienced SCA to determine if there is a genetic basis for SCA.

DETAILED DESCRIPTION:
SCA occurs when the heart suddenly and unexpectedly stops beating. When this happens, blood stops flowing to the brain and other vital organs. Ninety-five percent of people who experience SCA die from it, most within minutes. SCA is usually caused by abnormal heart rhythms, known as arrhythmias, which can be triggered by several factors, including coronary artery disease, physical stress, and structural changes in the heart. Certain genetic factors may also increase the likelihood of experiencing SCA. Study researchers will analyze genetic samples from people affected by SCA and people unaffected by SCA to identify and characterize genetic variations that are associated with an increased risk of SCA in European Americans and African Americans.

This study will examine previously collected blood samples from people who have experienced SCA and were participants in the Cardiac Arrest Blood Study (CABS) and the Cardiovascular Health Study (CHS). These participants will not attend any study visits or be contacted by study researchers. People who experience SCA in the first 4 years of this study will have blood drawn from paramedics at the time of SCA. If these participants survive, they will be asked whether study researchers can review their medical records. Study researchers will also examine previously collected blood samples from participants who have not experienced SCA and were participants in CABS, CHS, and the Heart and Vascular Health Study. These participants will not attend any study visits or be contacted by study researchers. Study researchers will also enroll a new control group of people who have not experienced SCA. These participants will attend one study visit for blood collection and a medical record review.

ELIGIBILITY:
Inclusion Criteria for People with SCA:

* Experienced incident SCA

Inclusion Criteria for People without SCA:

* Matched to people with SCA on age, gender, and ethnicity

Exclusion Criteria for People with SCA and without SCA:

* Members of a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group of people who have experienced SCA will be selected from participants in the Cardiac Arrest Blood Study (CABS), participants in the Cardiovascular Health Study (CHS), and residents of Seattle and King County, WA who experience SCA.
  The control group of people who have not experienced SCA will be selected from participants in CABS, participants in the Heart and Vascular Health Study, participants in CHS, and residents of Seattle and King County, WA who have not experienced SCA.
Sampling Method: Non-Probability Sample
Enrollment: 14862 (Actual)
Dates: Start 2007-09; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Genetic factors that may predispose people to develop SCA | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Nona Sotoodehnia, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Cardiovascular Health Research Unit, University of Washington, Seattle, Washington, United States